CLINICAL TRIAL: NCT00121589
Title: Lutein/Zeaxanthin and Omega-3 Supplementation in Persons Over Age 60
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050073; 05-EI-0073
Record Dates: First submitted 2005-07-20; First posted 2005-07-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Macular Degeneration
Keywords: AMD; Macular Pigment; Serum Lutein Levels; Vitamin Supplementation; Carotenoids; Lutein; Zeaxanthin; DHA; Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein

INTERVENTIONS:
Drug: Lutein

SUMMARY:
This study will explore whether taking the vitamins lutein and zeaxanthin, with or without Omega-3 fatty acid (fish oil or docosahexanoic acid, also known as DHA) will change the amount of lutein and zeaxanthin in the blood among people with age-related macular degeneration (AMD). AMD is one of the leading causes of legal blindness among people over the age of 50 in developed countries. In the disease, the retina of the eye, the sensory portion, worsens in condition. AMD causes progressive loss of central vision, with only peripheral vision remaining, that is, the ability for someone to see from the edges of the eye. To date, there is not any effective treatment to improve vision for most people whose AMD is advanced. Yet some data from research studies suggest a possible role of antioxidants, including lutein, in reducing the risk of AMD and cataracts. Lutein and zeaxanthin belong to the carotenoid family of vitamins, of which there are more than 600. There are 40 or 50 carotenoids in the typical diet of human beings, but only 14 major dietary ones are identified in human plasma. Lutein, in particular, is a vitamin that is found naturally in the retina, especially in the macula, the region of the eye that is essential for fine, detailed vision. Previous studies have shown that higher levels of foods rich in Omega-3 fatty acid were associated with a lower likelihood of AMD.

Patients ages 60 and older who may or may not have AMD, who do not have certain other serious eye disorders, and who have not had potentially life-threatening illness in the last year may be eligible for this study. About 40 people will participate.

Patients will undergo a medical history and physical examination. A blood collection of about 4 tablespoons will be done to measure the amount of lutein and other vitamins in the blood. Patients will have a complete eye examination consisting of procedures standard to those given by ophthalmologists. Participants will have photographs taken of their eyes, and they will undergo a visual field test. Flicker photometry also will be conducted. This consists of the patients looking at a flashing bluish light with one eye at a time, and turning a knob until the light stops flashing. Then during the test, patients will look away from the light and turn the knob until the flashing stops.

During this study study, patients will be asked to not take more than two tablets each day of multivitamins that contain lutein. The vitamin supplements will be provided as pills that represent one of two vitamin regimens given on a random basis: either lutein and zeaxanthin with DHA or lutein and zeaxanthin without DHA added. The amounts would be 10 mg/day of lutein and 2 mg/day of zeaxanthin, with or without 1 g/day of DHA. Patients will return to the study center for follow-up visits at 1 month, 3 months, 6 months, and 9 months. During those visits, some of the examinations done earlier will be repeated so that the researchers can evaluate the effects of supplements on patients' eyes. Patients will also be watched for possible side effects from the vitamins supplements. Lutein and zeaxanthin supplements are considered to be safe with possible minor side effects, such as headaches and difficulty in swallowing the tablets. Fish oil or DHA supplements may also cause abdominal discomfort.

If information obtained from this study may be important for participants' health, they will be informed when it is available. There are no plans to give participants the results of any medical tests, evaluations, or other research data. Further research may be necessary before such results become meaningful.

DETAILED DESCRIPTION:
The current proposed study is a necessary pilot study to prepare for a large-scale phase III randomized clinical trial planned to investigate whether oral supplementation with macular xanthophylls (lutein and zeaxanthin) and omega-3 long-chain polyunsaturated fatty acids (LCPUFAs) will decrease the progression of age-related macular degeneration (AMD) when compared to placebo. The primary objective of this pilot study is to investigate whether additional oral supplementation of omega-3 LCPUFAs (1 g/day) to daily supplementation of lutein (10 mg/day) and zeaxanthin (2 mg/day) will change the plasma levels of lutein and zeaxanthin in participants over age 60. The secondary objective is to study whether changes in serum levels of xanthophylls, lutein and zeaxanthin following oral supplementation will result in changes in the macular pigment density. In this study, forty participants (20 participants per arm) will take the study medications of lutein (10 mg/day) and zeaxanthin (2 mg/day) with or without the omega-3 LCPUFAs (1 g/day) for 6 months and will be followed for a total of 9 months (the initial 6 months with supplementation and the last 3 months without supplementation). Participants will range from those with no AMD and little or no drusen in either eye through advanced AMD (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in one eye. AMD severity will be classified using Age-Related Eye Disease Study (AREDS) criteria for the definition of advanced AMD. This is a preliminary study to be conducted prior to a large-scale phase III randomized clinical trial of omega -3 LCPUFAs and lutein/zeaxanthin for patients with moderate to high risk of AMD. The estimates of increases in serum lutein and zeaxanthin levels and the corresponding changes of macular pigment densities will provide essential information in conducting a large phase III randomized trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will range from those with no AMD and little or no drusen in either eye through end stage AMD (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in one eye. AMD severity will be classified using AREDS criteria for the definition of advanced AMD. Children are not included because AMD is, by definition, an adult disease and the study is designed to assess the effect of oral administration of lutein in persons in the age group affected by AMD.

* Men and women aged 60 years or older.
* Eligible participants may have no evidence of AMD with little or no drusen in either eye, or may have any stage of AMD through end stage (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in one eye.
* The ability to understand and sign an informed consent form prior to enrollment.
* People who currently smoke are eligible to enroll in this study. However, if smokers take an AREDS-like supplement, they must not take the AREDS-like supplement during the study.

EXCLUSION CRITERIA:

* Ocular disease (other than AMD) which confounds assessment of the retina including diabetic retinopathy, central serous choroidopathy, optic atrophy, retinal vein occlusion, active uveitis, significant explained or unexplained visual field loss, or any other type of retinopathy or retinal degeneration.
* Chronic requirement for any systemic or ocular medication for other eye diseases such as glaucoma.
* Regular use of lutein/zeaxanthin of 6 mg or more: during the last 3 months or currently taking these supplements. The daily use of the new Centrum or Centrum Silver or other similar multivitamins will be allowed but is limited to a maximum of twice a day.
* Participant has regularly taken 1 gm of fish oil (DHA, EPA) during the last 3 months or currently taking fish oil supplementation
* Inability or unwillingness to be followed for the nine-month study period.
* Acute, potentially life-threatening illness such as heart attack in the last year, or malignancy or blood disease not in remission.
* Any history of lung cancer.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07-14; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bone RA, Landrum JT, Hime GW, Cains A, Zamor J. Stereochemistry of the human macular carotenoids. Invest Ophthalmol Vis Sci. 1993 May;34(6):2033-40. PMID 8491553